CLINICAL TRIAL: NCT05485844
Title: A Case-control Study Comparing Women With Increased Symptoms (Back Pain and Core Stability Problems) and Inter Rectus Diameter a Year After Index Pregnancy.
Brief Title: Low Back Pain and Motor Control Dysfunction After Pregnancy- the Possible Role of Abdominal Rectus Muscle Diastasis
Acronym: D2
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jaana Vironen, Associate Professor, Helsinki University Central Hospital
Other Study IDs: HUS/3331/2017
Record Dates: First submitted 2022-07-27; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Diastasis Recti

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic: Individuals reporting increased back pain and/or decreased motor control function in a second questionnaire conducted a year after index pregnancy
- Controls: Controls reporting no change in their bodily experience between the two questionnaires

SUMMARY:
The aim of this study was to compare participants with increased symptoms after index pregnancy with those reporting no change in back pain or subjective movement control and analyzed their inter rectus distance (IRD). This study is a case-control study of a cohort of women who had delivered a year earlier. We recruited participants with increased symptoms (n=14) after index pregnancy and controls (n=41) and recorded their inter rectus distance with ultrasound. A questionnaire was filled, and an ultrasound was performed two times for the study groups.

DETAILED DESCRIPTION:
A case control study was conducted in Helsinki University Hospital during 1.1.2018-31.3.2021.

Participants were enrolled in pregnancy screening unit. Exclusion criteria was pregnancy during the second questionnaire and body mass index over 28kg/m2. The first questionnaire was filled and the baseline width of linea alba was measured by abdominal ultrasound (US) in connection of the first early pregnancy screening during 1.1.2018-8.3.2019. The second electronic questionnaire was sent a year after the expected delivery timing. Two screening questions were used to grade the participants. Altogether 36 individuals scored at least five points reflecting to substantial increase in symptoms in screening questions in the second questionnaire after pregnancy out of which fourteen participants were randomly recruited. Another 94 individuals scored the lowest possible two points implicating no change in ones bodily experience. Three controls per case were recruited, altogether 42 controls and with one dropout the total number of controls was 41. All participants had at least 12 months from the last delivery.

Two physiotherapists conducted motor control tests and the width of linea alba was measured with a high-end ultrasound. The physiotherapists were blinded with group allocation and the previous IRD measurement. Participants did not know their own exposure status or their IRD when answering the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years

Exclusion Criteria:

* Body mass index (BMI) over 28 kg/m2 ( weight and height combined to report BMI in kg/m^2
* Ongoing pregnancy during the second questionnaire, a year after the index pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A study is for abdominal rectus diastasis after pregnancy
Study Population: Participants were enrolled in pregnancy screening unit during the first pregnancy screening ultra sound.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-21 (Actual)

PRIMARY OUTCOMES:
Inter rectus diameter | A year after index pregnancy
  Ultra sound measurement of linea alba widht

SECONDARY OUTCOMES:
Waiter's bow | A year after index pregnancy
  Lumbar flexion motor control test performed in a standardized manner, with dichotomous rating of correct and non-correct performance. Rating was performed by a blinded specialist of physiotherapy from video recording.
Pelvic tilt | A year after index pregnancy
  Lumbar extension motor control test performed in a standardized manner, with dichotomous rating of correct and non-correct performance. Rating was performed by a blinded specialist of physiotherapy from video recording.
One leg stance-test | A year after index pregnancy
  Postural and balance control control test performed in a standardized manner, with dichotomous rating of correct and non-correct performance. Rating was performed by a blinded specialist of physiotherapy from video recording.
Active straight leg test | A year after index pregnancy
  Lumbar spine stability and abdominal bracing ability test performed in a standardized manner, with dichotomous rating of correct and non-correct performance. Rating was performed by a blinded specialist of physiotherapy from video recording.
Sit up test | A year after index pregnancy
  Arms crossed in front of the chest, elbows touch the knees in upright position. Sole can rise from the floor only slightly so that the angle of the hip does not change. Performance was video recorded and rating was performed by a blinded specialist of physiotherapy.
RAND36 HRQoL | A year after index pregnancy
  RAND36 HRQoL survey each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Jorvi Hospital, Espoo, HUS, Finland

IPD SHARING:
Plan to Share IPD: No